CLINICAL TRIAL: NCT03978988
Title: Intracranial Thrombectomy and Extracranial Carotid Stenting Versus Intracranial Thrombectomy Alone In Acute Anterior Circulation Strokes With TANdem Occlusion : the Randomized Controlled TITAN Trial
Brief Title: Thrombectomy In TANdem Occlusion
Acronym: TITAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Benjamin GORY, MD, PhD, MD, PhD, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A01085-52
Record Dates: First submitted 2019-05-29; First posted 2019-06-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Carotid Artery Diseases; Thrombectomy; Tandem Occlusion; Stroke
Keywords: stroke; tandem occlusion; carotid stenting; thrombectomy
MeSH Terms: conditions — Carotid Artery Diseases; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Thrombectomy + Carotid Stenting (Experimental): Intravenous thrombolysis will be administered if possible. Standard mechanical thrombectomy(MT) will be performed with a balloon Guide Catheter. MT technique will be left at the discretion of the operators.
  Concerning the cervical disease, emergent carotid stenting will be performed if the patient is randomized in the intervention arm. The order to treat (head first or neck first), and the choice of a previous angioplasty of the extracranial carotid artery lesion will be left to the interventionist discretion. An intravenous bolus of 250mg of Aspirin (up to Imaging 24H) will be given at the end of the procedure in case of absence of complication.
  Intravenous sedation or general anesthesia will be permitted.A second antiplatelet agent is used if a thrombus is formed : IV or nasogastric tube (choice by operator) A dual antiplatelet therapy is administered after 24H imaging follow-up excluding intracranial hemorrhagic complications (discretion of the local practice)
  Interventions: Device: Carotid Stenting; Drug: Procedural Aspirin; Drug: Dual dual antiplatelet therapy after 24-hours imaging follow-up; Procedure: Intracranial thrombectomy
- Thrombectomy alone (No Intervention): Endovascular procedure:
  Intracranial thrombectomy alone (carotid angioplasty may be performed)

INTERVENTIONS:
Device: Carotid Stenting — emergent carotid stenting will be performed if the patient is randomized in the intervention arm. The order to treat (head first or neck first), and the choice of a previous angioplasty of the extracranial carotid artery lesion will be left to the interventionist discretion.
  Arms: Thrombectomy + Carotid Stenting
Drug: Procedural Aspirin — After carotid stenting, an intravenous bolus of 250mg of Aspirin will be given at the end of the procedure in case of absence of complication.
  Arms: Thrombectomy + Carotid Stenting
Drug: Dual dual antiplatelet therapy after 24-hours imaging follow-up — A dual antiplatelet therapy is administered after 24-hours imaging follow-up excluding intracranial hemorrhagic complications (the type and the dose of the dual antiplatelet therapy are left to the discretion of the local practice)
  Arms: Thrombectomy + Carotid Stenting
Procedure: Intracranial thrombectomy — Intracranial thrombectomy is the endovascular procedure. In the experimental group, thrombectomy will be completed with a extracranial carotid stenting.
  Arms: Thrombectomy + Carotid Stenting

SUMMARY:
Tandem occlusion is defined by an acute ischemic stroke (AIS) with concomitant steno-occlusive disease of the extra cranial carotid artery and concerned about 10% of AIS patients. Whereas endovascular treatment has shown its efficiency in AIS by large vessel occlusion (LVO), to date, there is no consensus on the endovascular management of the extra cranial carotid artery in tandem occlusion. Only few of them were included in previous randomized trials who evaluated mechanical thrombectomy and were often listed in the non-inclusion criteria. Therapeutic management of this population was not specifically addressed in recent trials. Endovascular management can be complex with the need of acute stenting of the extra cranial carotid lesion along with the potential need of antithrombotic therapy initiation, the benefit and the safety of stenting of the cervical lesion in acute phase of AIS have shown encouraging results but however remains to be assessed. The TITAN (Thrombectomy In TANdem lesion) trial aims to demonstrate the superiority of the combined use of intracranial thrombectomy and extracranial carotid stenting compared to intracranial thrombectomy alone on the complete reperfusion rate in patients with acute ischemic stroke due to tandem lesion.

DETAILED DESCRIPTION:
The TITAN trial is a prospective, randomized, multi center, controlled, open-label, blinded clinical trial. This academic trial designed to answer the question: "What is the best endovascular management of the extra cranial carotid artery lesion in tandem occlusion with LVO" Patients will be recruited at 13 comprehensive stroke centers in France, all of which regular conduct mechanical thrombectomy and carotid stenting.

This study will enroll adults patients admitted with cerebral infarction of the anterior circulation, proven by computed tomography (CT) or magnetic resonance (MR) angiography, associated with tandem lesion, within 8 hours of symptoms onset, with a neurological deficit NIHSS > 5, and eligible to thrombectomy according to the recommendations of the French societies of neurovascular disease and neuroradiology (SFNR and SFNV).

Tandem occlusion of the anterior circulation will be proven on digital subtraction angiography, defined as a proximal intracranial occlusion and an extracranial severe internal carotid artery (ICA) lesion (complete occlusion or stenosis ≥90% North American Symptomatic Carotid Endarterectomy Trial).

Informed Consent according to the French laws will be sought from the patient if their level of consciousness is sufficient or from a relative. This study will operate using an emergency inclusion protocol due to the nature of the condition.

After emergency inclusion procedure according to French regulations, eligible patients will be randomized in two balanced parallel groups to receive either combined treatment intracranial thrombectomy with carotid stenting or intracranial thrombectomy alone.

Treatment and Intervention Intravenous thrombolysis will be administered if possible. Standard MT will be performed with a balloon Guide Catheter (BGC). MT technique (contact aspiration, stent retriever, or solumbra) will be left at the discretion of the operators.

Concerning the cervical disease, emergent carotid stenting will be performed if the patient is randomized in the intervention arm. The order to treat (head first or neck first), and the choice of a previous angioplasty of the extracranial carotid artery lesion will be left to the interventionist discretion. An intravenous bolus of 250mg of Aspirin will be given at the end of the procedure in case of absence of complication. (Aspirin 250mg IV up to Imaging 24H).A second antiplatelet agent is used if a thrombus is formed : IV or nasogastric tube (choice by operator)

Primary objective :

To demonstrate the superiority of intracranial thrombectomy and extracranial carotid stenting compared to intracranial thrombectomy alone on the complete reperfusion (mTICI 3 at the end of the endovascular procedure) rate and on the rate of NIHSS ≥ 4 points improvement at 24 hours in AIS patients with a tandem occlusion of the anterior circulation.

Secondary objectives :

1. To assess the feasibility and the efficacy of the combined approach associating intracranial thrombectomy and extracranial carotid stenting compared to intracranial thrombectomy alone using a composite criterion (mTICI3 at the end of the endovascular procedure or NIHSS improvement ≥ 4 points at 24h).
2. To compare the safety of intracranial thrombectomy and extracranial carotid stenting compared to intracranial thrombectomy alone.
3. To evaluate the cost-effectiveness and cost-utility of the combined approach compared to intracranial thrombectomy alone.

The Data and Safety Monitored Board (DSMB) will provide subject safety oversight and make recommendations to the Sponsor regarding continuing enrollment, modifying, or stopping the study early based upon a review of safety data and more specifically the comparative rates of symptomatic intracranial hemorrhage and, neurological worsening (NIHSS4 points increase), at D1, and mortality rates. They will take into account in their decision making and recommendations the rates of procedure-related and device-related events in the treatment group.

DSMB meetings will be organized by call conference by the sponsor before the start of the study and every year until the end of the study. The members will also receive the results of interim analyses. Additional extraordinary meetings will be set if necessary.

It will be constituted with two independent clinicians and one expert in methodology.

Sample Size Estimates Prior data indicate that a reperfusion rate of 30% mTICI 3 was observed with mechanical thrombectomy in patients with tandem lesions. Assuming acute carotid stenting will bring a 15% gain, a sample size of 162 patients per group will allow to evidence such gain with a 80% power at a 5% type I error (PS v3.0). Allowing 5% loss to follow up leads to include 216 patients per group, i.e. 432 patients in total

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged ≥ 18 years
2. Tandem occlusion confirmed by MR angiography or CT-angiography or digital subtraction angiography of supra-aortic vessels, in connection with atheromatous plaque or dissection, defined with:

   * Proximal intracranial occlusion (ICA, M1 and/or M2) eligible for thrombectomy
   * Extracranial lesion of the internal carotid artery (stenosis ≥90% NASCET or complete occlusion).
3. NIHSS Score ≥ 6
4. Arterial puncture performed :

   -> Within 8 hours (after the first symptoms or last seen well) with ASPECTS Score ≥5 by CT or MRI (DWI)

   OR

   -> Between 8 and 24 hours :
   * If perfusion imaging performed: according to the DEFUSE3 trial criteria (ischemia ≤70 mL, ischemia-hypoperfusion ratio≥1.8, and hypoperfusion volume ≥15 mL)
   * If perfusion imaging not performed: according to the DAWN trial criteria :

     * Age ≥80 years with NIHSS ≥10 and ischemia ≤21 mL
     * Age <80 years with NIHSS ≥10 and ischemia ≤31 mL
     * Age <80 years with NIHSS ≥20 and ischemia ≤51 mL
5. The patient or his or her representative has received information about the study organization and has signed and dated the informed consent form/ inclusion in emergency situation in accordance with Article L1122-1-3 of the Public Health Code.
6. Person affiliated to or beneficiary of a social security plan
7. Person undergone the medical examination adapted to research Subjects treated with prior intravenous thrombolysis are eligible for participation

Exclusion Criteria:

1. Extracranial internal carotid artery stenosis < 90% (NASCET)
2. Rankin score (mRS) > 2
3. Contraindication to antiplatelet (Aspirin, Plavix), or thrombolytic therapy (Actilyse), or contrast agents, or endovascular products.
4. Patient unable to present or be available for follow-up
5. Patient's refusal to participate
6. Woman of childbearing age without effective contraception
7. Pregnant, parturient or breastfeeding woman
8. Minor person (non emancipated)
9. Adult person under legal protection (any form of public guardianship)
10. Person deprived of liberty for judicial or administrative decision
11. Person under psychiatric care according to articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Change in Modified treatment in cerebral ischemia (mTICI) score AND National Institutes of Health Stroke Scale (NIHSS) score | at the end of angiography(mTICI score) , at 24 hours (NIHSS score)
  Complete reperfusion rate at the end of angiography defined as a modified Thrombolysis in Cerebral Infarction (mTICI) 3 score and defined as an Improvement of the National Institutes of Health Stroke Scale (NIHSS) score ≥ 4 mTICI score : 0:no perfusion ; 1:penetration with minimal perfusion ; 2:partial perfusion
  ; 2a:partial filling of less than 1/2 of the vascular territory ; 2b:partial filling 50-99% of the vascular territory ; 3:complete perfusion .
  NIHSS : 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items.

SECONDARY OUTCOMES:
Efficacy outcomes : Rate of reperfusion with change in Modified treatment in cerebral ischemia (mTICI) score | at the end of the endovascular procedure
  Complete reperfusion rate at the end of angiography defined as a modified Thrombolysis in Cerebral Infarction (mTICI) 3 score.
  mTICI score (0,1,2,2a,2b,3) : Grade 0 : no perfusion Grade 1 : penetration with minimal perfusion Grade 2 : partial perfusion Grade 2a : partial filling of less than 1/2 of the vascular territory Grade 2b : partial filling 50-99% of the vascular territory Grade 3 : complete perfusion
Efficacy outcomes : Change in National Institutes of Health Stroke Scale (NIHSS) score | at 24 hours (±6) hours
  NIHSS improvement ≥ 4 points at 24 (±6) hours (blinded assessment : core laboratories of 2 independent neuroradiologists).
  National Institutes of Health Stroke Scale (NIHSS) score. The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The single patient assessment requires less than 10 minutes to complete. The evaluation of stroke severity depends upon the ability of the observer to accurately and consistently assess the patient.
Efficacy outcomes : number of participants with delays of symptoms | at the end of the endovascular procedure
  - Delays of symptoms onset to groin puncture, groin puncture to clot contact, groin puncture to reperfusion, and symptoms onset to reperfusion
Efficacy outcomes : Number of passes | at the end of the endovascular procedure
  Number of intracranial thrombectomy passes to achieve final reperfusion
Efficacy outcomes : Infarct growth (volume) | At 24hours (±6) hours
  Infarct growth difference between treatment and control groups expressed as difference in Alberta Stroke Program Early CT score (ASPECT scores) at 24 (±6) hours.
  ASPECT scores : A 10-point score to assess ischemic stroke in the territory of the middle cerebral artery on a brain scan without injection.
  Calculated on a CT without axial cross-sectional injection:
  No hypodensity = 1 point Score = 10: total absence of hypodensity Score = 0 : hypodensity of the entire middle cerebral artery (MCA)territory A score ≤7 = pejorative prognosis in terms of both residual disability and risk of haemorrhagic transformation
Efficacy outcomes : Type and dose of antiplatelet agents administered | at 24 (±6) hours, at discharge (5-7 days)
  Type and dose of antiplatelet agents administered during the procedure, at 24 (±6) hours, at discharge (5-7 days).
Efficacy outcomes : Rate of recurrent clinical ischemic event | at 90 days for rate of recurrent clinical ischemic event
  Rate of recurrent clinical ischemic event at 90 (±15) days in the ipsilateral carotid territory
Efficacy outcomes : Rate of functional independence | at 90 days and 12 months for mRS
  - Rate of functional independence defined as a modified Rankin Scale (mRS) score 0-2 at 90 (±15 days) and 12 months (blind and independent evaluation) The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. Standardized interviews to obtain a mRS score are recommended at 3 months (90 days) following hospital discharge.
Safety outcomes : Rate of procedural complications | At the end of endovascular procedure
  Rate of procedural complications: vascular perforation, arterial dissection, embolization to new territory, access site complication requiring surgical repair or blood transfusion, intra-procedural mortality, and device failure
Safety outcomes : Rates of carotid stenosis and stent thrombosis | At the end of endovascular procedure
  Rates of carotid stenosis and stent thrombosis at the end of the endovascular procedure
Safety outcomes : Rate of symptomatic and asymptomatic intracerebral hemorrhage | at 24 hours (±6 hours)
  Rate of symptomatic and asymptomatic intracerebral hemorrhage at CT (Computerized Tomography) or MRI (Magnetic Resonance Imaging) at 24 hours (±6 hours) according to the Heidelberg classification (independent imaging core laboratory)
Safety outcomes : Rate of carotid stenosis and stent thrombosis | at 24 (±6) hours
  Rate of carotid stenosis (NASCET : North American Symptomatic Carotid Endarterectomy Trial Collaborators), and stent thrombosis at 24 (±6) hours on Computerized Tomography Angiography (CTA) or Magnetic Resonance Angiography (MRA)
Safety outcomes :Rate of secondary decompressive craniotomy | at discharge (or 5-7 days)
  Rate of secondary decompressive craniotomy at discharge (5-7 days)
Safety outcomes : Rate of endarterectomy | at 90 days and 12 (±1) months
  Rate of endarterectomy at 90 (±15) days, and 12 (±1) months
Safety outcomes : Rate of mortality | at 24 (±6) hours, 90 (±15) days, and 12 (±1) months
  Rate of mortality at 24 (±6) hours, 90 (±15) days, and 12 (±1) months
Cost effectiveness outcomes : value the additional cost of gaining additional clinical (NIHSS) | At 24 hours
  A cost-effectiveness analysis on secondary outcome criteria will be conducted to value the additional cost of gaining additional clinical benefit at 24 hours (NIHSS), and at 3 months (mRS), especially in terms of functional ability, using an incremental cost-effectiveness ratio. The result will be presented as cost per additional case of disability averted.
Cost effectiveness outcomes : value the additional cost of gaining additional clinical (mRS) | at 3 months
  A cost-effectiveness analysis on secondary outcome criteria will be conducted to value the additional cost of gaining additional clinical benefit at 24 hours (NIHSS), and at 3 months (mRS), especially in terms of functional ability, using an incremental cost-effectiveness ratio. The result will be presented as cost per additional case of disability averted.
Cost effectiveness outcomes : cost of safety issues | At 3 months
  Cost of safety issues will be considered. The time horizon will be at 3 months. The analysis will be conducted in the National Health Insurance System (NHIS) perspective. For this purpose, the investigators will classify each patient's stay in the appropriate Diagnosis-Related Group (DRG).
Cost effectiveness outcomes : a cost-utility analysis | At 12 months
  in a perspective of generic comparison, a cost-utility analysis will be conducted by using quality of life scores collected at 12 months of the intervention. The objective is to estimate the cost by one quality-adjusted life year (QALY) gained.
Cost effectiveness outcomes : a budget impact analysis | At 12 months
  a budget impact analysis will be performed. The objective is to estimate the total cost of adopting the combined approach of treatment at the national level and the expected number of disability cases averted.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin GORY, PhD, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Zhu F, Hossu G, Soudant M, Richard S, Achit H, Beguinet M, Costalat V, Arquizan C, Consoli A, Lapergue B, Rouchaud A, Macian-Montoro F, Biondi A, Moulin T, Marnat G, Sibon I, Paya C, Vannier S, Cognard C, Viguier A, Mazighi M, Obadia M, Hassen WB, Turc G, Clarencon F, Samson Y, Dumas-Duport B, Preterre C, Barbier C, Boulanger M, Janot K, Annan M, Bricout N, Henon H, Soize S, Moulin S, Labeyrie MA, Reiner P, Pop R, Wolff V, Ognard J, Timsit S, Reyre A, Perot C, Papagiannaki C, Triquenot-Bagan A, Bracard S, Anxionnat R, Derelle AL, Tonnelet R, Liao L, Schmitt E, Planel S, Guillemin F, Gory B. Effect of emergent carotid stenting during endovascular therapy for acute anterior circulation stroke patients with tandem occlusion: A multicenter, randomized, clinical trial (TITAN) protocol. Int J Stroke. 2021 Apr;16(3):342-348. doi: 10.1177/1747493020929948. Epub 2020 Jun 9. PMID 32515696